CLINICAL TRIAL: NCT02529397
Title: Obesity Treatment Enhanced With Working Memory Training
Acronym: Focus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Jean R. Harvey, PhD, RD, Professor and Chair, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHRBBS: 15-647
Record Dates: First submitted 2015-08-18; First posted 2015-08-20 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: ADHD; Weight Loss
Keywords: Working Memory Training, Weight Loss,
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adaptive Working Memory Training (Experimental): The experimental group will receive working memory training through a commercial computerized program: five weeks of adaptive working memory training concurrently with a behavioral weight loss program. Adaptive working memory training becomes progressively more challenging depending on an individual's performance on a given task. They will attend weekly classes of a behavioral weight loss program.
  Interventions: Behavioral: Adaptive Working Memory Training
- Non-adaptive Working Memory Training (Placebo Comparator): The control group will receive five weeks of non-adaptive (placebo) cognitive training concurrent with the identical behavioral weight loss program as in the experimental group. Non-adaptive cognitive training remains at a constant level.
  Interventions: Behavioral: Non-adaptive cognitive training

INTERVENTIONS:
Behavioral: Adaptive Working Memory Training — Participants will train for 30-40 minutes per day, five days per week at home for 5 weeks using an adaptive cognitive training program which becomes increasingly challenging as the participant masters each level. Behavioral classes will teach the principles of weight management and exercise.
  Arms: Adaptive Working Memory Training
Behavioral: Non-adaptive cognitive training — Participants will train for 30-40 minutes per day, five days per week at home for 5 weeks using a non-adaptive cognitive training program. Behavioral classes will teach the principles of weight management and exercise.
  Arms: Non-adaptive Working Memory Training

SUMMARY:
This study will examine the effects of providing subjects who have attention deficits, with or without a formal diagnosis of attention deficit hyperactivity disorder (ADHD), with Working Memory computerized training and explore whether this training is a feasible way to help them better engage in a weight loss treatment program, thereby enhancing weight loss results. Half of the participants will receive five weeks of online adaptive WM training concurrently while attending an in-person 24-week behavioral weight management program and half will receive five weeks of a non-adaptive form of cognitive training concurrently while attending a 24-week behavioral weight management program in person.

DETAILED DESCRIPTION:
Populations with ADHD or attention issues tend to have more weight loss attempts, struggle more with losing weight, and drop out of treatment more frequently than those without attention difficulties. Adaptive working memory training has been used to strengthen working memory and to mediate the symptoms associated with ADHD. The adaptive training becomes progressively more challenging as participants master each level of the training, while non-adaptive training remains at the same level throughout. Both groups will attend 24 weekly, in-person weight management classes on the University of Vermont Campus. Both groups will do cognitive training on their own home computers five days a week for 30-40 minutes for five weeks concurrently while engaged in the weight loss program.

ELIGIBILITY:
Inclusion Criteria:

* Must score 4 or higher on the ASRS v. 1.1
* Must live within 45 minutes driving distance from UVM campus
* Must be able to exercise
* Must have a computer with internet access and ability to utilize flash
* Must be 18 or older

Exclusion Criteria:

* Health issues that preclude exercise
* use of medications that interfere with the ability to lose weight
* vacation longer than two weeks
* current participation in another weight loss program
* reside more than 45 minutes from UVM campus in Burlington
* no internet access, no home computer, or computer cannot use flash

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Weight | 24 weeks
  Participants weight at baseline will be compared to their weight at 24 weeks at the completion of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Doris Ogden, MS, Principal Investigator — University of Vermont
Locations (1):
- Behavioral Weight Management Program/Univ of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Undecided